CLINICAL TRIAL: NCT01688349
Title: Comparative Study of Subcutaneous and Visceral Adipose Tissue in Patients Affected by Cushing Syndrome Versus 2 Controls Population
Brief Title: Pattern of Gene Expression in Adipose Tissue From Patients With Cushing Syndrome
Acronym: LIPOCUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P110906; CRC11001 (Other: Assistance Publique)
Record Dates: First submitted 2012-08-02; First posted 2012-09-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Cushing Syndrome Related to Cortisolic Adenoma
Keywords: Glucocorticoids; adipose tissue; Cushing; lipodystrophy; 11 beta-HSD1
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cushing group (Experimental): AT biopsy during partial nephrectomy
  Interventions: Other: analyze the role of glucocorticoid in AT distribution.
- Controls1 (Other): normal weight metabolic healthy patients having partial nephrectomy with small AT Biopsy.
  Interventions: Other: analyze the role of glucocorticoid in AT distribution.
- Controls2 (Other): obese individuals already included and having biopsies of VAT and SCAT stocked.
  Interventions: Other: analyze the role of glucocorticoid in AT distribution.

INTERVENTIONS:
Other: analyze the role of glucocorticoid in AT distribution. — The purpose of this trial is to investigate the impact of cortisol on adipose tissue functions, distribution and morphology. Patient with endogenous blood cortisol excess exhibit changes in adipose tissue, with fat gain in the upper trunk, face and neck leading to visceral obesity and features of the metabolic syndrome. The aims of this study will be
  * to compare the pattern of gene expression between visceral and subcutaneous adipose tissue in Cushing patients requiring an adrenalectomy as cortisol adenoma treatment;
  * to compare these patterns of gene expression with those of two control populations:1/ healthy metabolic subjects having a partial nephrectomy, 2/obese patients with similar degree of insulin resistance.

SUMMARY:
The purpose of this trial is to investigate the impact of cortisol on adipose tissue functions, distribution and morphology. Patient with endogenous blood cortisol excess exhibit changes in adipose tissue, with fat gain in the upper trunk, face and neck leading to visceral obesity and features of the metabolic syndrome. The aims of this study will be

* to compare the pattern of gene expression between visceral and subcutaneous adipose tissue in Cushing patients requiring an adrenalectomy as cortisol adenoma treatment;
* to compare these patterns of gene expression with those of two control populations:1/ healthy metabolic subjects having a partial nephrectomy, 2/obese patients with similar degree of insulin resistance.

DETAILED DESCRIPTION:
Cushing's syndrome is a rare disease resulting from chronic exposure to glucocorticoids (endogenous or iatrogenic) with abnormal fat distribution (lipodystrophy). Glucocorticoids regulate the functions of adipose tissue (AT) targeting adipocyte differentiation as well as anabolic, catabolic and secretory pathways of the adipocyte. However, the mechanisms by which glucocorticoids differentially disrupt the development or metabolism of AT between deep and superficial deposits remain unknown. Among the main effectors of the glucocorticoid signaling pathway, 11 beta-hydroxysteroid deshydrogenase (11beta-HSD1) , that regenerate cortisol from cortisone, is likely a key step in the biological effect of glucocorticoids in AT. Identifying these mechanisms of action of glucocorticoids on different fat depots requires the comparison with fatty deposits derived from two types of control populations: 1/ normal weight individuals without inflammatory or metabolic disorder (controls1); 2/individuals obese matched for the level of insulin resistance (controls2).

Hypothesis: Excess glucocorticoids cause abnormal fat distribution via a direct effect on the various deposits of AT, leading secondarily to insulin resistance.

Primary endpoint: To compare gene expression of glucocorticoid signaling between the visceral AT (VAT) of Cushing patients with that of controls1 (matched for age and sex).

Secondary endpoints:

1. For patients with Cushing and controls1, to compare their respective subcutaneous AT (SCAT) and VAT for:

   * The expression of genes involved in differentiation and inflammation of the AT,
   * Morphological aspects: adipocyte size, fibrosis, inflammation, immunohistochemistry.
2. Same parameters for Cushing patients and controls2 (matched for sex, age + / -5, HOMA-R + / -1), to differentiate the specific effects of glucocorticoid from the effects of insulin resistance,
3. To compare these parameters between SCAT and VAT from Cushing patients. Methodology and experimental design: non-randomized comparative multicenter study with constitution of a biological collection.

Patients will be recruited in endocrinology before adrenalectomy and controls1 in urology. They will have a preoperative assessment and sampling of perirenal AT and SCAT at surgery. Controls2 are already included in the CRC2007-P050318 and will be drawn for matching.

Number of patients needed: We assume the relative gene expression of 11β-HSD1 in the VAT not exposed to glucocorticoids = 0.81 ± 0.121. Our recruitment potential of Cushing patients is 30 patients. With 30 patients per group, we will be able to detect a difference in 11β-HSD1 gene expression in the VAT of Cushing patients at least 15% higher compared to controls1.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Adults with Cushing's syndrome secondary to adrenal adenoma.
* Controls1: Adults with normal weight: BMI <25, having partial nephrectomy
* Controls2 adults with common obesity treated by bariatric surgery, BMI> 35kg/m2

Exclusion Criteria:

* Diabetes, renal or hepatic impairment, pregnancy, menopause, HIV or HCV, Cushing's syndrome due to other causes than cortisol adenoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

PRIMARY OUTCOMES:
Comparison between visceral adipose tissue of Cushing patients and that of normal weight controls. | 1 day (gene expression will be tested on AT withdraw the day of surgical adrenalectomy)
  Comparison of glucocorticoid pathway genes expression between visceral adipose tissue of Cushing patients and that of normal weight controls matched on sex and age.

SECONDARY OUTCOMES:
Comparison of the respective SCAT and VAT between Cushing patients and normal weight controls. | 1 day (gene expression will be tested on AT withdraw the day of surgical adrenalectomy)
  For patients with Cushing and controls1, to compare their respective SCAT and VAT for:
  * The expression of genes involved in differentiation and inflammation of the AT,
  * Morphological aspects: adipocyte size, fibrosis, inflammation, immunohistochemistry.
Comparison of the respective SCAT and VAT between Cushing patients and obese controls. | 1 day (gene expression will be tested on AT withdraw the day of surgical adrenalectomy)
  Comparison of these same parameters(secondary outcome n°1) between Cushing patients and controls2 (matched for sex, age + / -5, HOMA-R + / -1), to differentiate the specific effects of glucocorticoid from the effects of insulin resistance
comparison between SCAT and VAT from Cushing patients | 1 day (gene expression will be tested on AT withdraw the day of surgical adrenalectomy)
  To compare these parameters between SCAT and VAT from Cushing patients

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Feve, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Hôpital Saint-Antoine, service d'Endocrinologie, Paris, France